Models of Care in the Transition from the Secondary to the Primary Sector among the Frailest Elderly +75; a Randomized Controlled Trial

Troels Kjærskov Hansen
Aarhus University Hospital
Randers Regional Hospital
Aarhus University
February 8th, 2019

# Models of Care in the Transition from the Secondary to the Primary Sector among the Frailest Elderly +75; a Randomized Controlled Trial

In most Western countries the elderly population increases rapidly. In Denmark, the population of elderly aged 75 years or older may amount to nearly 15 % of the entire population in 2050 compared to 9 % today (2017) (1). A large part of the elderly population is at high risk of hospitalization including more admissions and increased morbidity and mortality (2,3). The number of hospital beds is declining persistently (4), calling for shorter lengths of stay (LOS) (5,6). Increasingly complex treatments now take place outside hospital. Presently, many Danish regional hospitals establish geriatric wards and other geriatric in-hospital and outpatient services to overcome these challenges. The aim of the present PhD-study is to investigate the effects of different models of transitional care among the frailest elderly patients.

#### Readmission

Readmitted patients occupy many beds and other hospital resources. Patients are at a risk of high mortality (7) and decline of functional ability (8,9). More than 20 % of Danish medical patients aged 65 years or older become readmitted within 30 days after discharge (10), more frequently in the frail elderly (11). The risk of readmission is particularly high within the first week after discharge, where more than 40% of readmissions happen (12,13). Many reasons and factors for readmissions have been mentioned (11,14-16) such as: former or recent admission, duration of the index hospitalization, degree of comorbidity and low functional ability (11,15). To prevent readmissions it is important to identify the reason for admission and remove it, to ensure that the correct medication is implemented and make sure that adequate social service is provided, to convey unsolved problems to the primary care, ensure continuity during transfer and finally establish sufficient and timely follow-up after discharge (11,14-17).

## Identification of patients at risk

Many factors leading to readmission and other adverse events are related to frailty (11,15,18). Prevention of adverse events has traditionally relied on clinicians' and caregivers' ability to anticipate the needs and requirements after discharge. Comprehensive Geriatric Assessment (CGA) is considered as the gold standard to detect frailty (19). To make this easier tools to determine frailty have been developed. In the present study the Multidimensional Prognostic Index (MPI; see Appendix 1A and 1B (slightly adjusted Danish version)) has been chosen to determine the level of frailty. MPI is fully applicable in the everyday clinical work and supplies useful information to clinicians, it is validated in a Danish context, predicts readmission and death (20), and is well-suited to assess the degree of frailty (18,21).

### Usual care

Present usual care in Denmark with regard to discharge and transfer, consists of discharge planning. It relies largely on the GP's follow-up visits (see Appendix 2). This approach reduces readmission (22), but the use is limited due to poor implementation, lack of referral, and missing follow-up despite referral (23,24). Only a minor fraction of the frail receives a follow-up visit within the first week after discharge. The GP-based intervention is presently subject to discussion (23,24). Urgent or hospital-at-home-like treatment is needed to avoid readmission. This requires of a well-informed round the clock service. The urgency of follow-up of the frail elderly does not fit into the scheme-based workday of the GP and the on-call GP system. In some districts, additional specialized geriatric wards and outgoing teams exist, but the capacity and contents of these units are limited and vary. Community nurses might after some reorganization hold an untapped potential to improve transition.

#### Counteractions to readmission

Even though all possible precautions are made before discharge, readmissions still occur. They are often preceded by a series of events stressing the need for multifaceted care and intersectoral efforts in relation to discharge. Many approaches are already applied:

- To avoid obvious and predictable events leading to readmission, comprehensive discharge planning has been introduced in many different countries, probably reducing readmission and LOS without increasing mortality (25,26).
- In a Danish context discharge follow-up is largely based on GP-conducted visits within one week after discharge and offered to a fraction of the elderly.
- Multiple discharge support arrangements have been tested ranging from isolated follow-up telephone calls by a hospital nurse to highly specialized multidisciplinary geriatric teams doing home visits. Early follow-up visits by community nurses have been tested showing possible effect on mortality but not on readmissions (27). Another recent randomized clinical trial (RCT) reports considerable positive effect on readmission, LOS and direct discharge from the ED (12), while a second RCT performed in the same population shows a reduction of

- mortality among patients living in their own homes (7). The study shows considerable effect of early team-based home visits applied on selected elderly at high risk of readmission (12).
- Comprehensive Geriatric Assessment (CGA) provides an individualized, multidisciplinary and intersectoral approach when applied by geriatricians in inpatient geriatric wards and in Emergency Departments (ED) and outpatient clinics, in order to improve outcomes of hospitalization. The effects of CGA on readmission, length of stay (LOS) or mortality has yet not been well-proven. It reduces medication and increases the probability of discharge at home (25,28). The effect of CGA combined with an early geriatric home visit has resulted in a significant reduction of the readmission rate within 30 days when compared to the GP-conducted follow-up visits after a week (12).

#### **Outcome measures**

According to the various interventions stated above, the outcomes of relevance are readmissions (8-12,15,17,22,24-26,28-44), mortality (7,8,10,12,25,27,28,30-32,38-41,44), length of stay (LOS) (12,25,28,29,32,38,41,45), direct discharge from the ED (12,29), time at home (10,25,27,34), duration of readmission (10,25,34) and physical functional status (8,25,27,28,30,31,34,40,43-45). A successful intervention may be reflected in a shorter LOS, lower risk of readmissions, longer time at home, maintained functional status and a shorter duration of readmission. We suggest that a significant and effective intervention under the best circumstances is reflected in these outcomes. Readmissions are usually considered as such, when the admission occurs within 4 hours after and before 30 days after discharge. Among the frail, in-hospital and post-discharge mortality is high, needing frequent assessment. As shown by Pedersen et al. (7), mortality differs with regard to type of dwelling. Former studies have shown a significant and remarkable reduction of LOS (reduction from median 3 days to median 2 days) and an increase from 49 % to 56 % of patients discharged directly from the ED due to the possibility of early follow up by a geriatric team (12). Functional status is of relevance, especially combined with mortality data, since a better survival of the frailest may be combined with a worsened functional status in the total group. Patient Related Outcome Measures (PROMs) will be assessed and added as secondary outcomes during the project. Patient satisfaction and costs are other relevant outcome measures with regards to the triple aim principle, but will not be included in the present Ph.D. project.

#### Conclusion

While some previously tested interventions, including CGA and discharge support arrangements, have been futile (25,31,46), we believe that multidisciplinary, tailored interventions used in selected high-risk groups throughout hospitalization and discharge are effective (8,12,29,34,44). Most former studies regarding early follow-up visits and CGA are made in geriatric settings, somewhat distanced to usual care and municipality services. Many previous trials have included patients without looking in particular for frail high-risk patients, thereby probably underestimating the effects of the intervention. It is not known if an early visit by a community nurse would have the same effect as an early geriatric home visit. Selection of elderly patients who will benefit from home visits by a geriatric team after discharge compared with a community nurse visit or usual care may be useful. MPI has been able to predict mortality, LOS (47), and readmissions (48), but has not previously been tested as a selection tool to distinguish between different follow-up methods. It has been suggested that the major effect from early follow-up is more or less independent of the type of follow-up, but is caused by the early visit itself. The type of dwelling may influence the effect of an early visit, since the care setup in some nursing homes may resemble that of a hospital. The level of frailty may influence the effectiveness and efficacy of the different follow-up schemes. Some patients may be chronically frail and their frailty may already have been handled prior to admission, in a way that dilutes the effect of early follow-up visits. The length of stay and other secondary endpoints may rely largely on the planned follow-up approach. The level of frailty predicts the risk of readmission and mortality and can therefore be used as a major indicator when clinicians have to choose between different follow-up approaches.

## **Objectives**

The aim of this study is to investigate the effects of two interventions using CGA and early post-discharge follow-up visits in a population of frail 75+ year-olds compared to usual care. The vision is to find feasible and durable approaches that can improve patient outcome in the transition from hospital to primary health care. We are aiming to identify subjects who will profit the most from each approach.

All frail patients admitted to the ED and the Department of Geriatrics are randomized 1:1 to one of two different follow-up efforts prior to CGA performed during hospitalization. Thereby the intervention is randomly split into two groups:

- An intervention (I) consisting of CGA during hospitalization and early post-discharge follow-up care by a community nurse and a GP
- An intervention (II) consisting of CGA during hospitalization and early post-discharge follow-up care, including continued CGA and tailored follow-up care, by a geriatric team

The intervention cohort will be compared to a control cohort consisting of similar frail elderly who receive usual care without involvement of geriatric care during hospitalization and after discharge.

## **Hypotheses**

- The geriatric team follow-up is as effective as a community nurse and GP follow-up measured by readmission, mortality, LOS, direct discharge from ED and physical functional recovery
- The effects of three transitional follow-up approaches (community nurse and GP; multidisciplinary geriatric team; usual care) are similar measured in terms of readmission, time at home, duration of readmission, LOS, direct discharge from ED, mortality and PROMs
- When stratified into subgroups with regards to level of frailty (moderate and severe) and type of dwelling, the geriatric team follow up is as good as community nurse and GP follow-up measured by readmission, mortality, LOS, direct discharge from ED and physical functional recovery

## **Methods**

## Design

The first study is conducted as a randomized controlled trial (RCT) using two different degrees of intervention. The second study is a cohort study where the two groups in the RCT are compared to an unexposed control group. The third study is sub-group analyses of the RCT data according to frailty status and type of dwelling.

## Study population

The population allocated to intervention comprises geriatric patients acutely admitted to the ED, Aarhus University Hospital (AUH) or transferred to one of the two geriatric wards at AUH. Subjects are included immediately on the day of admission at the ED, AUH and the Department of Geriatrics (wards 1 and 2), AUH, as shown in Fig. 1. Patients admitted to the ED at night and promptly discharged before enrollment to the intervention cohort can be performed the following day are not included. Likewise, patients to the control group are included immediately on the day of admission at the ED, Randers Regional Hospital (RRH), and at the medical wards 1, 2, 3 and 4, RRH. Patients transferred to other departments are excluded. Patients can only be included once. Enrollment and randomization to the intervention group are performed by therapists working in the ED or the geriatric wards. Enrollment to the control group is done by a Research Assistant. In the control group frailty screening is done by the PhD-student using a frailty screening tool based exclusively on data collected through medical records. The frailty screening tool will be validated by crosschecks performed by a blinded project Research Assistant. The results of the validation study will be analyzed and published during 2019.

#### **Inclusion criteria:**

- Aged 75 years or older
- Living within the municipality of Aarhus (except for the control group, see below)
- MPI-score = 2 (moderate frailty) or MPI score = 3 (severe frailty)

### **Exclusion criteria:**

- Included in any other kind of follow-up schemes
- Declared terminally ill or undergoing palliative care at admission
- Admitted from one specific temporary nursing home with geriatric medical assistance (Vikærgården)
- Discharge or transfer to another department, including hospice
- MPI-score = 1 (low frailty)
- Discharged to one specific temporary nursing home with geriatric medical assistance (Vikærgården)
- The patient does not want a visit after discharge

Inclusion- and exclusion criteria to the control group are the same as for the two intervention groups, except that subjects eligible for the control group are living within the four municipalities of RRH: Randers, Favrskov, Norddjurs and Syddjurs.

#### Randomization

As shown in Fig. 2, all intervention group patients are allocated at the time of randomization on the day of admission to receive either early visit from the community nurse (I) or the multidisciplinary geriatric team (II). The randomization is stratified with regard to dwelling (living alone; cohabiting; nursing home) and number of drugs prescribed prior to

admission (0-3, 4-7, 8 or more drugs), and conducted using the randomization function in REDCap (49). Randomization is open throughout the whole admission with the purpose to enable early discharge planning.

#### Intervention I and II

Both intervention groups are assessed according to CGA, either by the geriatrician and the physiotherapist/geriatric nurse in the ED, or by a multidisciplinary team comprised of geriatricians, specialized nurses, physiotherapists and occupational therapists during hospitalization in the geriatric wards.

- Intervention (I): comprises early follow-up visit from the community nurse within 24 hours after discharge, and the possibility of consulting a nutritionist, thus supplementing usual care services including the possibility of consulting the patients' GP. Responsibility of treatment including implementation of suggested initiatives and any further assessment is handed over to the GP at discharge.
- Intervention (II): CGA is continued during early follow-up by the geriatric team. On weekdays visits are scheduled within 24 hours after discharge. For patients discharged during weekends or holidays, supporting telephone calls are provided by the geriatric team. If needed, the geriatric team nurse visits the patient. The concept of CGA in this stage does not differ from the above-mentioned. There are no standardized demands, but a part of the intervention can be to perform hospital services at home and continued treatment and diagnostics after discharge. The possible services provided by the geriatric team are further described in the geriatric team course description. The responsibility of treatment rests with the geriatric team until dispatch of the discharge summary. Patients then return to usual care. The geriatric team follow-up is planned to last a maximum of 7 days, yet allowing extension for as long as there is a need for services performed exclusively by the geriatric team as described in the geriatric team course description.

### Control group

The patients in the control group are discharged to usual care and do not receive early follow-up visits. Usual care features municipality services and optionally a GP home visit (see Appendix 2). Eligible control patients are consecutively included by a Research Assistant. The estimated level of frailty will be assessed by the PhD-student based on a MPI-screening tool fitted to be performed using only medical record data. This fitted tool will be tested and validated prior to the inclusion of the control group. Clinicians will be blinded to the result of the MPI-screening of the control subjects to ensure that discharge is performed in accordance with usual care.

## **Outcomes**

The primary outcome is readmission within 30 days after discharge. Secondary outcomes are:

- Mortality 30 days after discharge and 90 days after admission
- Length of stay during primary admission and total length of stay including following readmissions
- Direct discharge from the Emergency Department
- Time at home before readmission
- Duration of readmission
- Physical functional status 30 days after discharge (Functional Recovery Score)
- Patient Related Outcome Measures as defined by a focus group of included patients and/or their relatives

## Statistical analyses

Data are registered in REDCap and exported to STATA version 15 for the statistical analyses. Statistical significant results are defined as a p-value of 5% or less. The two intervention groups and the control group will be compared with regard to baseline measures. If needed, statistical corrections for demographical differences and level of frailty will be made. The use of services and other contents of follow-up will be assessed and compared if possible. Baseline data collected for the entire study population before discharge are: age, gender, date of admission, co-habitation status, number of drugs, and level of frailty measured by MPI including functional status by means of Functional Recovery Score (FRS) at discharge. Follow-up data for the control group will be collected on type of planned care after discharge. Follow-up data for the entire study population will be collected on: department of discharge, date of discharge, primary diagnosis at discharge, dwelling after discharge, readmission date, and death date. For the intervention cohort additional data are collected: date of follow-up, provided services after discharge, number and date of visits (team, GP, nurse) after discharge, phone-calls to the geriatric team or GP, nutritionist consultations, FRS after 30 days, date of dispatch of discharge summary. Additional data will be collected by review of the electronic patient records.

#### Outcomes

A hazard ratio (HR) for readmissions will be calculated using a Cox regression model with death as a 'competing risk' factor. The HRs of readmission with 95% confidence intervals (95% CI) for interventions I and II will be compared individually and to the control group. The interventions will be tested in subgroup analyzes based on: patients discharged directly from the ED, type of dwelling and level of frailty. Median LOS, time at home before readmission and duration of readmission will be calculated and compared using the Wilcoxon rank-sum test. The mortality hazard ratio will be calculated also using the Cox regression model. The change in functional status at discharge and 30 days after discharge will be compared in a linear regression model. Data will be analyzed in accordance with intention-to-treat and perprotocol analysis.

#### Sample size

Power analysis is based on a pilot study performed from June to December 2017 using the method stated above, and earlier studies by Pedersen et al.(7,12), where patients selected by diagnoses associated with readmission were randomized to early geriatric follow-up visits or usual care. Readmissions were reduced from 23% to 12%. Data collected during the pilot study showed 13.7% readmissions in the Intervention group I compared to 8% readmissions in the Intervention group II. Based on the pilot study data, allowing a 5% drop-out rate and a 30-day mortality rate of 10%, the number of patients in each trial arm should be 758 in order to achieve a power of 90% and a level of significance of 5%. Data collected during the same pilot study showed a 90-day mortality rate of 20.6% in Intervention group I compared to 15.6 % in Intervention group II. To achieve a power of 80% and a level of significance of 5% with regards to mortality, the sample size of each arm should be 1,019, including a 5% drop-out rate.

## **Perspectives**

This study may uncover a need for specialized and early efforts to support transfer of the frail elderly. We may find that some of the frail elderly are poorly supported by the present follow-up procedures, suggesting that comprehensive geriatric assessment and early follow-up intervention by a community nurse and a geriatric team should gain further currency in the future. This study may contribute to dimension health care services in the future. We hope to clarify the possible need for geriatric services outside university hospitals. The results are directly transferable to Danish regional hospitals and may be of importance in other Western countries.

#### Ethics

The study has been approved as a quality development project by the Regional Research Ethics Committee, Central Denmark Region (journal no. 197/2017), thereby no patient consent form is needed, and further referral to the committee not required. No patient will receive less than usual care, no extra treatment or examination will be applied, and no patient will be exposed to any additional risk because of the project. Participants may decline parts of or the entire intervention, including usual care, at any time. The project, which is a part of the national rate adjustment pool-project "Early post-discharge follow-up of the frail elderly – a intersectoral effort" in the Central Denmark Region, is approved by the Danish Data Protection Agency (journal no. 2012-58-006).

# Organization and economy

The project is embedded in the Geriatric Department, Aarhus University Hospital. The project is conducted in cooperation with Aarhus Municipality, represented by health consultant, PhD, Monica Milter Ehlers, and Randers Regional Hospital, where professor, MD, PhD, Jens Meldgaard Bruun and MD, geriatric specialist, Seham Shahla will be co-supervisors. See Fig. 3. The Project Manager, MD, PhD-student Troels Kjærskov Hansen, will be employed at both hospitals as a clinical assistant. The day-to-day work will take place mainly in the Research Unit at the Geriatric Department, AUH under supervision of the main supervisor, professor, MD, PhD, Else Marie Damsgaard, and co-supervisor, clinical specialist, PhD, Merete Gregersen. Through the Geriatric Department, AUH, there will be available statistical expertise attached to the project. Data regarding the intervention group will be collected by the research assistants associated to the Geriatric Department, AUH with regard to the frailty screening and baseline characteristics. Functional status at follow-up will be assessed by Aarhus municipality research assistants. The three months' leave for writing the project protocol was sponsored by the Central Denmark Region's Health Research Foundation. Follow-up as well as the hospital and municipality research assistants are partly funded by the Rate Adjustment Pool, the Geriatric Department, AUH, and Aarhus Municipality. Future expenses will be PhD student salary, Study Fee, wage for a research assistant, costs of courses, congresses, transportation, and publication.

# My part

The Project Manager is admitted to the PhD programme and PhD courses at Aarhus University. The PhD-student is responsible for the collection, storage, analysis and correctness of all data. The PhD-student will apply for the remaining funding and publish and present the data from the project in relevant peer-reviewed journals and at national and international congresses. The project is reported to ClinicalTrials.gov. Research Plan: see Appendix 3.

## References

- (1) Danmarks Statistik. Statistikbanken. Available at: www.dst.dk. Accessed 1009, 2017.
- (2) Sundhedsdatastyrelsen. Ældre medicinske patienters kontakt med det regionale sundhedsvæsen og den kommunale pleje. 2016; Available at: <a href="https://sundhedsdatastyrelsen.dk/da/nyheder/2016/aeldre-medicinske-patienter-sundhedsvæsen\_14042016">https://sundhedsdatastyrelsen.dk/da/nyheder/2016/aeldre-medicinske-patienter-sundhedsvæsen\_14042016</a>. Accessed September, 2017.
- (3) Danmarks Statistik. Sygehusbenyttelse 2015. 2015; Available at: http://www.dst.dk/Site/Dst/Udgivelser/nyt/GetPdf.aspx?cid=23069. Accessed September, 2017.
- (4) Sundhedsdatastyrelsen. Sengepladser fordelt på specialer 1996-2013. 2013; Available at: <a href="http://esundhed.dk/sundhedsaktivitet/SOB/Sider/SOB02.aspx">http://esundhed.dk/sundhedsaktivitet/SOB/Sider/SOB02.aspx</a>. Accessed September, 2017.
- (5) Kommunernes Landsforening KL. Udvikling i gennemsnitlig indlæggelsestid blandt unge, voksne og ældre fra 2008 til 2013. 2015; Available at: <a href="http://www.kl.dk/ImageVaultFiles/id">http://www.kl.dk/ImageVaultFiles/id</a> 74350/cf 202/Analyse af udvikling i indl-ggelsestid.PDF. Accessed September, 2017.
- (6) Kommunernes Landsforening KL. Udvikling i indlæggelsesvarighed for somatiske indlæggelser. 2017; Available at: <a href="http://www.kl.dk/ImageVaultFiles/id\_83744/cf\_202/Udvikling\_i\_indl-ggelsesvarighed\_for\_somatiske\_ind.PDF">http://www.kl.dk/ImageVaultFiles/id\_83744/cf\_202/Udvikling\_i\_indl-ggelsesvarighed\_for\_somatiske\_ind.PDF</a>. Accessed September, 2017.
- (7) Pedersen LH, Gregersen M, Barat I, Damsgaard EM. Early geriatric follow-up after discharge reduces mortality among patients living in their own home. A randomised controlled trial. Eur Geriatr Med 2017 2017/09;8(4):330-336.
- (8) Caplan GA, Williams AJ, Daly B, Abraham K. A randomized, controlled trial of comprehensive geriatric assessment and multidisciplinary intervention after discharge of elderly from the emergency department The DEED II study. J Am Geriatr Soc 2004 /;52(9):1417-1423.
- (9) Pedersen MK, Meyer G, Uhrenfeldt L. Risk factors for acute care hospital readmission in older persons in Western countries: a systematic review. JBI DATABASE SYST REV IMPLEMENT REP 2017 02;15(2):454-485.
- (10) Pedersen MK, Nielsen GL, Uhrenfeldt L, Rasmussen OS, Lundbye-Christensen S. Description of OPRA: A Danish database designed for the analyses of risk factors associated with 30-day hospital readmission of people aged 65+ years. Scand J Public Health 2017 08;45(6):595-604.
- (11) Benbassat J, Taragin M. Hospital readmissions as a measure of quality of health care: Advantages and limitations. Arch Intern Med 2000 2000/04;160(8):1074-1081.
- (12) Pedersen LH, Gregersen M, Barat I, Damsgaard EM. Early geriatric follow-up after discharge reduces readmissions A quasi-randomised controlled trial. Eur Geriatr Med 2016 2016/09;7(5):443-448.
- (13) Ministeriet for Sundhed og Forebyggelse. Forebyggelse af indlæggelser synlige resultater. 2014; Available at: <a href="http://www.sum.dk/~/media/Filer%20-%20Publikationer\_i\_pdf/2014/Forebyggelse-af-indlaeggelser-synlige-resultater-maj-2014/Forebyggelse-af-indlaeggelser-synlige-resultater-maj-2014.ashx.">http://www.sum.dk/~/media/Filer%20-%20Publikationer\_i\_pdf/2014/Forebyggelse-af-indlaeggelser-synlige-resultater-maj-2014/Forebyggelse-af-indlaeggelser-synlige-resultater-maj-2014.ashx.</a> Accessed October, 2017.
- (14) Forster AJ, Murff HJ, Peterson JF, Gandhi TK, Bates DW. The incidence and severity of adverse events affecting patients after discharge from the hospital. Ann Intern Med 2003 2003/02;138(3):161-167.
- (15) García-Pérez L, Linertová R, Lorenzo-Riera A, Vázquez-Díaz JR, Duque-González B, Sarría-Santamera A. Risk factors for hospital readmissions in elderly patients: A systematic review. QJM 2011 /;104(8):639-651.
- (16) Naylor MD, Shaid EC, Carpenter D, Gass B, Levine C, Li J, et al. Components of Comprehensive and Effective Transitional Care. J Am Geriatr Soc 2017 2017/06;65(6):1119-1125.
- (17) Scott IA. Preventing the rebound: Improving care transition in hospital discharge processes. Aust Health Rev 2010 /:34(4):445-451.

- (18) Dent E, Kowal P, Hoogendijk EO. Frailty measurement in research and clinical practice: A review. Eur J Intern Med 2016 2016/06;31:3-10.
- (19) Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet 2013 /;381(9868):752-762.
- (20) Gregersen M, Hansen TK, Jørgensen BB, Damsgaard EM. Validation of a modified Multidimensional Prognostic Index obtained at discharge in older Danish geriatric patients to predict acute readmission and mortality. 2018 Unpublished data.
- (21) Warnier RMJ, van Rossum E, van Velthuijsen E, Mulder WJ, Schols JMGA, Kempen GIJM. Validity, reliability and feasibility of tools to identify frail older patients in inpatient hospital care: A systematic review. J Nutr Health Aging 2016 2016/02;20(2):218-230.
- (22) Rytter L, Jakobsen HN, Rønholt F, Hammer AV, Andreasen AH, Nissen A, et al. Comprehensive discharge follow-up in patients' homes by GPs and district nurses of elderly patients. A randomized controlled trial. Scand J Prim Health Care 2010/;28(3):146-153.
- (23) Hendriksen C, Vass M. Uncertain efficiency of follow-up home visits among older patients after hospital discharge. Ugeskr Laeg 2014 2014/01;176(5):V04130264.
- (24) Thygesen LC, Fokdal S, Gjørup T, Taylor RS, Zwisler A-. Can municipality-based post-discharge follow-up visits including a general practitioner reduce early readmission among the fragile elderly (65+ years old)? A randomized controlled trial. Scand J Prim Health Care 2015 2015/06;33(2):65-73.
- (25) Parker SG, Peet SM, McPherson A, Cannaby AM, Abrams K, Baker R, et al. A systematic review of discharge arrangements for older people. Health Technol Assess 2002 2002/;6(4).
- (26) Dedhia P, Kravet S, Bulger J, Hinson T, Sridharan A, Kolodner K, et al. A quality improvement intervention to facilitate the transition of older adults from three hospitals back to their homes. J Am Geriatr Soc 2009 /;57(9):1540-1546.
- (27) Buurman BM, Parlevliet JL, Allore HG, Blok W, Van Deelen BAJ, Moll Van Charante EP, et al. Comprehensive geriatric assessment and transitional care in acutely hospitalized patients the transitional care bridge randomized clinical trial. JAMA Intern Med 2016 2016/03;176(3):302-309.
- (28) Ellis G, Gardner M, Tsiachristas A, Langhorne P, Burke O, Harwood RH, et al. Comprehensive geriatric assessment for older adults admitted to hospital. Cochrane Database Syst Rev 2017 2017/09;2017(9).
- (29) Conroy SP, Ansari K, Williams M, Laithwaite E, Teasdale B, Dawson J, et al. A controlled evaluation of comprehensive geriatric assessment in the emergency department: The 'Emergency Frailty Unit'. Age Ageing 2014 /;43(1):109-114.
- (30) Kircher TTJ, Wormstall H, Müller PH, Schwärzler F, Buchkremer G, Wild K, et al. A randomised trial of a geriatric evaluation and management consultation services in frail hospitalised patients. Age Ageing 2007 /:36(1):36-42.
- (31) Conroy SP, Stevens T, Parker SG, Gladman JRF. A systematic review of comprehensive geriatric assessment to improve outcomes for frail older people being rapidly discharged from acute hospital: 'Interface geriatrics'. Age Ageing 2011 /;40(4):436-443.
- (32) Gregersen M, Pedersen ABL, Damsgaard EM. Comprehensive geriatric assessment increases 30-day survival in the aged acute medical inpatients. Dan Med J 2012 2012/;59(6).
- (33) Oates DJ, Kornetsky D, Winter MR, Silliman RA, Caruso LB, Sharbaugh ME, et al. Minimizing Geriatric Rehospitalizations: A Successful Model. Am J Med Qual 2013 /;28(1):8-15.
- (34) Naylor MD, Brooten D, Campbell R, Jacobsen BS, Mezey MD, Pauly MV, et al. Comprehensive discharge planning and home follow-up of hospitalized elders: A randomized clinical trial. J Am Med Assoc 1999 1999/02;281(7):613-620.

- (35) Linertová R, García-Pérez L, Vázquez-Díaz JR, Lorenzo-Riera A, Sarría-Santamera A. Interventions to reduce hospital readmissions in the elderly. Value Health 2010 /;13(7):A406.
- (36) Shen E, Koyama SY, Huynh DN, Watson HL, Mittman B, Kanter MH, et al. Association of a dedicated post-hospital discharge follow-up visit and 30-day readmission risk in a Medicare advantage population. JAMA Intern Med 2017 2017/01;177(1):132-135.
- (37) Huntley AL, Chalder M, Shaw ARG, Hollingworth W, Metcalfe C, Benger JR, et al. A systematic review to identify and assess the effectiveness of alternatives for people over the age of 65 who are at risk of potentially avoidable hospital admission. BMJ Open 2017 2017/07;7(7).
- (38) Gonçalves-Bradley DC, Iliffe S, Doll HA, Broad J, Gladman J, Langhorne P, et al. Early discharge hospital at home. Cochrane Database Syst Rev 2017 2017/06;2017(6).
- (39) Altfeld SJ, Shier GE, Rooney M, Johnson TJ, Golden RL, Karavolos K, et al. Effects of an enhanced discharge planning intervention for hospitalized older adults: a randomized trial. Gerontologist 2013 /;53(3):430-440.
- (40) Nikolaus T, Specht-Leible N, Bach M, Oster P, Schlierf G. A randomized trial of comprehensive geriatric assessment and home intervention in the care of hospitalized patients. Age Ageing 1999 1999/;28(6):543-550.
- (41) Shepperd S, Iliffe S, Doll HA, Clarke MJ, Kalra L, Wilson AD, et al. Admission avoidance hospital at home. Cochrane Database Syst Rev 2016 2016/09;2016(9).
- (42) Coleman EA, Parry C, Chalmers S, Min S-. The care transitions intervention: Results of a randomized controlled trial. Arch Intern Med 2006 2006/09;166(17):1822-1828.
- (43) Harris R, Ashton T, Broad J, Connolly G, Richmond D. The effectiveness, acceptability and costs of a hospital-athome service compared with acute hospital care: A randomized controlled trial. J Health Serv Res Policy 2005 /;10(3):158-166.
- (44) Naylor MD, Brooten DA, Campbell RL, Maislin G, McCauley KM, Schwartz JS. Transitional Care of Older Adults Hospitalized with Heart Failure: A Randomized, Controlled Trial. J Am Geriatr Soc 2004 /;52(5):675-684.
- (45) Mas MA, Inzitari M, Sabate S, Santaeugenia SJ, Miralles R. Hospital-at-home Integrated Care Programme for the management of disabling health crises in older patients: comparison with bed-based Intermediate Care. Age Ageing 2017 Nov 1;46(6):925-931.
- (46) Linertová R, García-Pérez L, Vázquez-Díaz JR, Lorenzo-Riera A, Sarría-Santamera A. Interventions to reduce hospital readmissions in the elderly: In-hospital or home care. A systematic review. J Eval Clin Pract 2011 /;17(6):1167-1175.
- (47) Volpato S, Bazzano S, Fontana A, Ferrucci L, Pilotto A. Multidimensional Prognostic Index predicts mortality and length of stay during hospitalization in the older patients: a multicenter prospective study. J Gerontol A Biol Sci Med Sci 2015 2015/03;70(3):325-331.
- (48) Daragjati J, Topinkova E, Puntoni M, Cruz-Jentoft A, Polidori MC, Paccalin M, et al. Multidimensional prognostic index (MPI) predicts re-hospitalization in frail older patients admitted to hospital: A multicentre, international, one-year follow-up study. the MPI-AGE European project. Eur Geriatr Med 2017 2017/09;8:S78-S79.
- (49) Vanderbilt University. REDCap. Available at: <a href="https://www.project-redcap.org/">https://www.project-redcap.org/</a>. Accessed November, 2017.



# REGIONE DEL VENETO AZIENDA ULSS 16 PADOVA

# OSPEDALE S. ANTONIO Unità Operativa Complessa di GERIATRIA

# MULTIDIMENSIONAL PROGNOSTIC INDEX (MPI) \*

## **CO-HABITATION STATUS**

| Does the patient live: |
|------------------------|
| Alone |
| With relatives/nourse |
| In institution |

# **MEDICATION USE**

| Number of drugs used |
|----------------------|

<sup>\*</sup> Pilotto A, Ferrucci L, Franceschi M et al. Development and validation of a Multidimensional Prognostic Index for 1-Year Mortality from a Comprehensive Geriatric Assessment in Hospitalized Older Patients. Rejuvenation Res 2008;11:151-161.

# ACTIVITIES OF DAILY LIVING (ADL) \*

| A) <b>BATHING</b> (either sponge bath, tub bath, or shower) | |
|---|---|
| - Receives no assistance (gets in and out of tub by self if tub is usual means of bathing) | 1 |
| - Receives assistance in bathing only one part of the body (such as back or a leg) | 1 |
| - Receives assistance in bathing more than one part of the body (or not bathed) | 0 |
| B) <b>DRESSING</b> (gets clothes from closets and drawers – including underclothes, outer garments, and using | |
| fasteners including braces, if worn) | |
| - Gets clothes and gets completely dressed without assistance | 1 |
| - Gets clothes and gets dressed without assistance except for assistance in tying shoes | 1 |
| - Receives assistance in getting clothes or in getting dressed, or stays partly or completely undressed | 0 |
| C) <b>TOILETING</b> (going to the "toilet room" for bowel and urine elimination, cleaning self after elimination | 1, |
| and arranging clothes) | |
| - Goes to "toilet room," cleans self, and arranges clothes without assistance (may use object for | 1 |
| support such as cane, walker, or wheelchair and may manage night bedpan or commode, | |
| emptying same in morning) | |
| - Receives assistance in going to "toilet room" or in cleaning self or in arranging clothes after | 0 |
| elimination or in use of night bedpan or commode | _ |
| - Doesn't go to room termed "toilet" for the elimination process | 0 |
| D) TRANSFER | 1 |
| - Moves in and out of bed as well as in and out of chair without assistance (may be using object | 1 |
| for support such as cane or walker) | _ |
| - Moves in and out of bed or chair with assistance | 0 |
| - Doesn't get out of bed | 0 |
| E) CONTINENCE | |
| - Controls urination and bowel movement completely by self | 1 |
| - Has occasional "accidents" | 0 |
| - Supervision helps keep urine or bowel control, catheter is used, or is incontinent | 0 |
| F) FEEDING | |
| - Feeds self without assistance | 1 |
| - Feeds self except for getting assistance in cutting meat or buttering bread | 1 |
| - Receives assistance in feeding or is fed partly or completely by using tubes or intravenous fluids | 0 |

| <b>TOTAL</b> |
|--------------|

<sup>\*</sup> Katz S, Ford AB, Moskowitz RW et al. Studies of illness in the aged. The index of ADL: A standardized measure of biological and psychological function. JAMA 1963; 185: 914-19.

# INSTRUMENTAL ACTIVITIES OF DAILY LIVING SCALE (IADL)\*

| A) ABILITY TO USE TELEPHONE | |
|---|---|
| - Operates telephone on own initiative: looks up and dials numbers, etc. | 1 |
| - Dials a few well-known numbers | 1 |
| - Answers telephone but does not dial | 1 |
| - Does not use telephone at all | 0 |
| B) SHOPPING | |
| - Takes care of all shopping needs independently | 1 |
| - Shops independently for small purchases | 0 |
| - Needs to be accompanied on any shopping trip | 0 |
| - Completely unable to shop | 0 |
| C) FOOD PREPARATION | • |
| - Plans, prepares and serves adequate meals independently | 1 |
| - Prepares adequate meals if supplied with ingredients | 0 |
| - Heats, serves and prepares meals or prepares meals but does not maintain adequate diet | 0 |
| - Needs to have meals prepared and served | 0 |
| D) HOUSEKEEPING | • |
| - Maintains house alone or with occasional assistance (e.g. "heavy work domestic help") | 1 |
| - Performs light daily tasks such as dishwashing, bed making, etc. | 1 |
| - Performs light daily tasks but cannot maintain acceptable level of cleanliness | 1 |
| - Needs help with all home maintenance tasks | 0 |
| - Does not participate in any housekeeping tasks | 0 |
| E) LAUNDRY | |
| - Does personal laundry completely | 1 |
| - Launders small items; rinses stockings, etc. | 1 |
| - All laundry must be done by others | 0 |
| F) MODE OF TRANSPORTATION | |
| - Travels independently on public transportation or drives own car | 1 |
| - Arranges own travel via taxi, but does not otherwise use public transportation | 1 |
| - Travels on public transportation when accompanied by another | 1 |
| - Travel limited to taxi or automobile with assistance of another | 0 |
| - Does not travel at all | 0 |
| G) RESPOSIBILITY FOR OWN MEDICTIONS | • |
| - Is responsible for taking medication in correct dosages at correct time | 1 |
| - Takes responsibility if medication is prepared in advance in separate dosage | 0 |
| - Is not capable of dispensing own medication | 0 |
| H) ABILITY TO HANDLE FINANCES | |
| - Manages financial matters independently (budgets, writes checks, pays rent, bills goes to bank), collects and keeps track of income | 1 |
| - Manages day-to-day purchases, but needs help with banking, major purchases, etc. | 1 |
| - Manages day-to-day purchases, but needs neip with banking, major purchases, etc Incapable if handling money | 0 |
| - incapable it nationing money | U |

| TOTAL |
|-------|
| IVIAL |

<sup>\*</sup> Lawton MP, Brody EM. Assessment of older people:self-maintaining and instrumental activities of daily living. Gerontologist 1969;9:179-86.

# SHORT PORTABLE MENTAL STATUS QUESTIONNAIRE (SPMSQ) \*

(Record the errors)

| What is the date today? (Correct only when the month, date, and year are all correct) | 1 |
|---|---|
| What day of the week is it? | 1 |
| What is the name of this place? (Correct if any of the description of the location is given) | 1 |
| What is your street address? | 1 |
| How old are you? | 1 |
| When were you born? | 1 |
| Who is the president (or the Pope) now? (Requires only the correct last name) | 1 |
| Who was president (or the Pope) just before him? | 1 |
| What was your mother's maiden name? | 1 |
| Subtract 3 from 20 and keep subtracting 3 from each new number at least for 3 times (The entire | 1 |
| series must be performed correctly to be scored as correct) | |

| <b>TOTAL</b> |
|--------------|
|--------------|

# **EXTON-SMITH SCALE (ESS) \***

(evaluation of pressure sores risk)

| General Condition | | Incontinence | |
|---|---|---|---|
| Bad Poor Fair Good Mental State | 1 Doubly incontinent 1 2 Usually of urine 2 3 Occasional 3 4 Not 4 4 | | |
| Stuporosous Confused Apathetic Alert | 3 | Immobile Very limited Slightly limited | 3 |
| Activity In bed all day Chairfast Walks with help Ambulant | 1 | Score 16-20: minimum risk | |

<sup>\*</sup> Bliss MR., McLaren R., Exton-Smith AN. Mattresses for preventing pressure sores in geriatric patients. Mon Bull Minist Health Public Health Lab Serv 1966

<sup>\*</sup> Pfeiffer E. A short portable mental status questionnaire for the assessment of organic brain deficit in elderly patients. J Am Geriatr Soc. 1975; 23:433-441.

# CUMULATIVE ILLNESS RATING SCALE (C.I.R.S.) \*

| | NONE | MILD | MODERATE | SEVERE | EXTREMELY<br>SEVERE |
|---|---|---|---|---|---|
| 1. Cardiac (heart only) | 1 | 2 | 3 | 4 | 5 |
| <b>2.</b> Hypertension (rating is based on severity) | 1 | 2 | 3 | 4 | 5 |
| 3. Vascular (arteries, veins, lymphatics) | 1 | 2 | 3 | 4 | 5 |
| 4. Respiratory (lungs, bronchi, trachea) | 1 | 2 | 3 | 4 | 5 |
| <b>5.</b> EENT (eye, ear, nose, throat, larynx) | 1 | 2 | 3 | 4 | 5 |
| <b>6.</b> Upper GI (esophagus, stomach, duodenum, biliary and pancreatic trees) | 1 | 2 | 3 | 4 | 5 |
| 7. Lower GI (intestines, hernias) | 1 | 2 | 3 | 4 | 5 |
| 8. Hepatic (liver only) | 1 | 2 | 3 | 4 | 5 |
| 9. Renal (kidneys only) | 1 | 2 | 3 | 4 | 5 |
| 10. Other GU (ureters, bladder, urethra, prostate, genitals) | 1 | 2 | 3 | 4 | 5 |
| 11. Musculo-skeletal-integumentary (muscles, bone, skin) | 1 | 2 | 3 | 4 | 5 |
| <b>12.</b> Neurological (brain, spinal cord, nerves) | 1 | 2 | 3 | 4 | 5 |
| <b>13.</b> Endocrine-metabolic (including diabetes, hyperlipidemia, infections, toxicity) | 1 | 2 | 3 | 4 | 5 |
| <b>14.</b> Psychiatric (dementia, depression, anxiety, agitation, psychosis) | 1 | 2 | 3 | 4 | 5 |

| ILLNESS SEVERITY SCORE (CIRS-IS) | COMORBIDITY INDEX (CIRS-CI) |
|---|---|
| mean of all single item | number of items with a score |
| (excluded the psychiatric item) | of 3 or greater (excluded the psychiatric item) |

<sup>\*</sup> Conwell Y, Forbes NT, Cox C, Caine ED. Validation of a measure of physical illness burden at autopsy: the Cumulative Illness Rating Scale. J Am Geriatr Soc 1993; 41: 38-41.

# MINI NUTRITIONAL ASSESSMENT (MNA) \*

A) Anthropometric Assessment 1) Body Mass Index (BMI) Weight: BMI < 19 BMI = 19-20BMI = 21-22 $BMI \ge 23$ Height: 2) Mid-arm circumference 0 0.5 MAC > 22(MAC) in cm MAC<21  $MAC \le 22$ 3) Calf circumference (CC) in cm CC < 31  $CC \ge 31$ 4) Weight loss 0 2 3 (last three months) loss > 3Kgdoes not know loss between 1-3Kg no weight loss B) General Assessment 5) Lives independently (not in a nursing home or hospital) 0 1 no yes 6) Takes more than 3 prescription drugs per day 0 1 yes no 7) Has suffered psychological stress or acute disease in the past 3 months 2 0 yes no 8) Mobility 0 bed or chair bound able to get out of bed/chair but goes out does not go out 9) Neuropsychological problems severe dementia or mild dementia no psychological problems depression 10) Pressure sores or skin ulcers 0 yes no C) Dietary Assessment 11) How many full meals does the 0 2 patient eat daily? 1 meal 2 meals 3 meals 12) Consumes: at least 1 serving of dairy 2 or more servings of meat, fisk or poultry Points if: products (milk, cheese, legumes or eggs per week every day 1 ves 0 yogurt) per day 2 yes 0.5 yes no yes no yes 3 yes 1 13) Consumes 2 or more servings of fruits or 0 vegetables per day? no yes 14) Has food intake declined over the 0 past 3 months due to loss of appetite? severe loss of appetite moderate loss of appetite no loss of appetite 15) How much fluidi s consumed per 0.5 less than 5 glasses 5 to 9 glasses more than 9 glasses 16) Mode of feeding 0 self-feed with some with assistance self-feed without any difficulty problem D) Self Assessment 17) Do they view themselves a s 0 having nutritional problems? major malnutrition does not know no nutritional problems 18) In comparison with other 0.5 people of same age, how they not as good does not know as good better consider their health status? **TOTALE** (max 30 punti) **MALNUTRITION INDICATOR SCORE**:  $\geq 24$  = well-nourished, 17-23.5 = at risk of malnutrition, < 17 = malnourished

<sup>\*</sup> Vellas B et al. The Mini Nutritional Assessment (MNA) and its use in grading the nutritional state of elderly patients. Nutrition 1999; 15: 116-22.

| | N N | Non (18-50 years)<br>Mon (60-00 years) | 1.04 | 1,93 | 1.92 | 1.01 | 1.90 | 1.89 | 1.88<br>1.88 | 1.87 | 1.865 | 1.86<br>1.85 | 1.81 | 1.84<br>1.83 | 1.62 | 1.82 | 1.81<br>1.80 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Kore height (cm) | 6.5 | 64.5 | 64 | 63.5 | 63 | 62.5 | 42 | 61.5 | 61 | 60.5 | 60 | 59.5 | 59 | 58.5 | 58 |
| | N N | Waters (18-50 years)<br>Waters (50-90 years) | 1.89<br>1.86 | 1.88 | 1.875<br>1.84 | 1.87 | 1.86 | 1.85 | 1.84<br>1.81 | 1.82 | 1.62 | 1.78 | 1.80 | 1.79<br>1.76 | 1.78 | 1.77 | 1.76 |
| Normogram for | THOM | Mon (18-59 years)<br>Mon ( 60-90 years) | 1.35 | 1.79<br>1.76 | 1.78 | 1.77 | 1.76 | 1.75 | 1.74 | 1.71 | 1.72<br>1.70 | 1.71 | 1.705<br>1.68 | 1.76 | 1.89 | 1.68<br>1.65 | 1,67 |
| the calculation | | Knee beight (end) | 57.5 | 57 | 56.5 | 56 | 55.5 | 55 | 54.5 | 54 | 83.5 | 83 | 52.5 | 52 | 51.5 | 51 | 50.5 |
| of knee height | N N | Winner (18-59 years)<br>Winner (60-00 years) | 1.75 | 1.74<br>1.71 | 1.735 | 1.00 | 1.72 | 1.67 | 1.70 | 1.65 | 1.68 | 1.67<br>1.63 | 1.625 | 1.65 | 1,64 | 1.69 | 1.50 |
| | ğ. | Mon (1.5-59 years)<br>Mon (60-90 years) | 1.66 | 1.65 | 1.61 | 1.63 | 1.62 | 1.51 | 1.57 | 1.59 | 1.58 | 1.57<br>1.54 | 1.54 | 1.555 | 1.55 | 1.54 | 1.53 |
| | - | Keen beight (cm) | 50 | 49.5 | 49 | 40.5 | 48 | 47.5 | 47 | 44.5 | (46) | 45,5 | 45 | 44.5 | 44 | 43.5 | 43 |
| | BE | Winners (1.6-50 years)<br>Winners (60-50 years) | 1.61<br>1.58 | 1.00<br>1.57 | 1.58 | 1.565 | 1.58 | 1.57 | 156 | 1.55 | 1.54 | 1.53 | 1.52 | 1.51 | 1.50 | 1.49 | 1.48 |

# **MPI - Multidimensional Prognostic Index**

| | Score given to each domain | | | | |
|---|---|---|---|---|---|
| | Low<br>(Value = 0) | Middl<br>(Value = | - | Hiç<br>(Value | |
| SPMSQ <sup>a</sup> | 0-3 | 4-7 | | 8-10 | |
| ESS <sup>b</sup> | 16-20 | 10-15 | | 5-9 | |
| ADL <sup>c</sup> | 6-5 | 4-3 | | 2-0 | |
| IADL <sup>c</sup> | 8-6 | 5-4 | | 3-0 | |
| CIRS d | 0 | 1-2 | | ≥ 3 | |
| MNA <sup>e</sup> | ≥ 24 | 17 to 23.5 | | <17 | |
| Number of drugs | 0-3 | 4-6 | | ≥ 7 | |
| Social status | Lives with family | Institutionalized | | Living | alone |
| Add up the scores as divide the sum by 8 | L SCORE | | | | |

Leaend:

| RISK Mild (MPI 1) | | Moderate (MPI 2) | Severe (MPI 3) |
|-------------------|-------------|------------------|----------------|
| RANGE | 0.00 - 0.33 | 0.34-0.66 | 0.67-1.0 |

to Number of errors

b Exton Smith Scale Score: 16-20, minimum risk, 10-15, moderate risk; 5-9, high risk of developing Number of active functional activities

d Number of pathological (score> 3)
e ≥ 24: satisfactory; 17-23.5: at risk of malnutrition; <17: Malnutrition

# Appendix 1B

(Slightly adjusted and translated (to Danish) version of Appendix 1A had to be removed since uploaded documents must be in English. If requested, Appendix 1B can be provided by the Record Owner Troels K. Hansen.)

# Usual post-discharge follow-up care

Usual care during transition comprises individualized discharge planning. In all cases, GPs receive an electronically transmitted discharge summary and an updated prescription list at discharge. Municipality services receive rehabilitation-and personal care plans and discharge reports made by hospital nurse. Post-discharge follow-up follows no fixed schedule or programme, thereby leaving assessment of care- and follow-up services to the municipality services, based on recommendations from hospital nurses and physicians. A variety of temporary and permanent nursing home facilities, rehabilitation units and other institutional living facilities exists.

Follow-up at home may include a visit by a community nurse and establishing or continuation of home care. Depending on screening during hospitalization, hospital nurses can by referral recommend a GP conducted home visit to patients aged 65 years or older. The actual execution of this home visit depends on the GPs judgment of its necessity. The screening process, leading to the proposal of a GP-conducted home visit, is based on data related to LOS, former admissions within the past year, functional status, state of nutrition, morbidity, medication, cognitive status, substance abuse, psychiatric diseases and coping ability. If the score is  $\geq 23$ , and the patient consents, the information is reported to the municipal health service and the GP. GPs may also on their own initiate a follow-up visit. The Danish College of General Practitioners recommends that the GP assesses the need for visit according to the following criteria:

- Health related issues: patients suffering from reduced functional or health related status prior to admission, need for assessment of medication, chronically and severely ill, impairment due to dementia, terminal illness.
- Organizational issues: patients readmitted, extended length of stay, need for assessment of coordinated efforts
- Social issues: frail and uneasy patients, weak social network, patients living alone, patients recently widowed If conducted, the home visit is performed within 8 days after discharge by the GP and/or community nurse. The contents of this intervention may be:
  - Evaluation of the discharge summary including changes of medication and specific follow-up needs specified.
  - Overall health assessment including functional status, for instance by means of chair stand test
  - Assessment of need for care and facilities
  - Medication review
  - Joint decision and plan

According to head nurses in the medical wards at Randers Regional Hospital, the screening and assessment of GP conducted follow-up visits is performed as a standard to all patients aged 65 years or older. Due to busyness, screening may sometimes be given low priority, particularly when knowing that many patients do not receive a visit despite referral. This is reflected in the recent data showing the numbers of screenings, number of referrals to and completion of visits (1).

# Appendix 3

| Year | | Jan | Feb | Mar | Apr | May | Jun | Jul | Aug | Sep | Oct | Nov | Dec |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 2017 | Pilot study MPI | | | | | Х | Х | Х | Х | Х | Х | | |
| | Writing protocol | | | | | | | | | Х | Х | Х | |
| | Randomization pilot | | | | | | | | | Χ | Х | Χ | |
| | MPI at discharge pilot | | | | | | | | | Χ | Χ | Х | |
| | Inclusion (Intervention) | | | | | | | | | | | Χ | Χ |
| 2018 | Inclusion (Intervention) | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Х | Х |
| | Writing article (method) | | | | | | | | | | | Х | X |
| 2019 | Validation study | Χ | Χ | Χ | | | | | | | | | |
| | Inclusion (Intervention) | Χ | Χ | Χ | Χ | Х | Χ | Χ | | | | | |
| | Inclusion (Control) | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| | PhD (until December 2021) | Х | Χ | Χ | Χ | Х | Х | Χ | Χ | Χ | Х | Χ | Χ |
| | Follow-up ends (Intervention) | | | | | | | | Χ | | | | |
| | Analyzing data (Intervention) | | | | | | | | Χ | Χ | Χ | Χ | Χ |
| | Writing articles | | | | | | Х | Χ | Χ | Χ | Χ | Χ | Χ |
| 2020 | Writing articles | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| | Follow-up ends (Control) | Х | | | | | | | | | | | |
| | Analyzing data (Control) | | Χ | Χ | Χ | Х | | | | | | | |
| | Writing PhD thesis | | | Χ | Х | Χ | Х | Х | Χ | Χ | Х | Χ | X |
| | 1 month abroad | | | | | | | | | | | Χ | X |
| 2021 | Writing PhD thesis | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | X |



# Randomization, discharge and follow-up



